CLINICAL TRIAL: NCT04912050
Title: EXtension of Tablo TrEatmeNt Duration Registry (XTEND)
Brief Title: EXtension of Tablo TrEatmeNt Duration Registry
Acronym: XTEND
Status: Completed | Type: Observational
Sponsor: Outset Medical (Industry)
Responsible Party: Sponsor
Other Study IDs: 2020-03
Record Dates: First submitted 2021-05-26; First posted 2021-06-03 (Actual); Last update posted 2022-08-12 (Actual); Status verified 2022-08

CONDITIONS: End Stage Renal Disease (ESRD); End Stage Renal Disease on Dialysis; Acute Kidney Injury
Keywords: Tablo; Outset Medical; Hemodialysis; AKI; ESKD
MeSH Terms: conditions — Kidney Failure, Chronic; Acute Kidney Injury

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Tablo Hemodialysis System: Hospitalized participants with End-Stage Kidney Disease or Acute Kidney Injury who are prescribed renal replacement therapy > 12 hours on the Tablo Hemodialysis System
  Interventions: Device: Tablo Hemodialysis System

INTERVENTIONS:
Device: Tablo Hemodialysis System — Renal Replacement Therapy between 12< to ≤ 24 hours.

SUMMARY:
Observational, retrospective and prospective, multicenter, post-market study of the Tablo Hemodialysis System in hospitalized participants with End-Stage Kidney Disease or Acute Kidney Injury who are prescribed renal replacement therapy > 12 hours.

ELIGIBILITY:
Inclusion Criteria:

* Participant weighs ≥ 34kg.
* Participant is hospitalized and has dialysis dependent End-Stage Kidney Disease or Acute Kidney Injury and is prescribed renal replacement therapy > 12 hours.

Exclusion Criteria:

* Any documented condition that the Physician feels would prevent the participant from successful inclusion in the study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Hospitalized participants with End-Stage Kidney Disease or Acute Kidney Injury who are prescribed renal replacement therapy > 12 hours.
Sampling Method: Non-Probability Sample
Enrollment: 33 (Actual)
Dates: Start 2021-05-25 (Actual); Primary Completion 2022-05-31 (Actual); Study Completion 2022-05-31 (Actual)

PRIMARY OUTCOMES:
Treatment Success | Up to 24 hours
  Percentage of treatments achieving prescribed dialysis treatment time ≤ 10%

SECONDARY OUTCOMES:
Tablo Cartridge Life | up to 24 hours
  Measure the average number of cartridge changes required to complete a Tablo XT Treatment

CONTACTS AND LOCATIONS:
Locations (1):
- St. Mark's Hospital, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: No
Only aggregated participant data is planned to be shared at this time.